CLINICAL TRIAL: NCT00338208
Title: Adult Providing Access to the Visual Environment (PAVE) - Glaucoma Pilot
Acronym: PAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Karen Joos, Associate Professor of Ophthalmology, Vanderbilt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vanderbilt IRB #030642
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Glaucoma
Keywords: low vision; glaucoma
MeSH Terms: conditions — Glaucoma; Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No training (No Intervention): Subjects will be fitted with low vision devices; no extra training will be provided.
- Training in the Use of Low Vision Devices (Experimental): Subjects will be fitted with low vision devices and will receive 6 training sessions with prescribed devices for up to 1 hour each time
  Interventions: Behavioral: Training in the Use of Low Vision Devices

INTERVENTIONS:
Behavioral: Training in the Use of Low Vision Devices
  Arms: Training in the Use of Low Vision Devices

SUMMARY:
We wish to evaluate a potential training program for patients with glaucoma, to become more efficient users of prescribed low vision devices for distance and near vision tasks. We hypothesize that the devices will improve efficiency. Prescribed devices will include a stand magnifier, a handheld magnifier, spectacle magnifiers for near vision, and a handheld monocular (telescope) and a bioptic telescope (spectacle-mounted telescope) for distance vision. The success of being able to use optical devices is dependent upon training. Optical devices are currently accepted and used for patients with visual conditions that decrease their central vision. The bioptic telescope is a pair of glasses with a small telescope mounted within the carrier lens. The glasses look and feel like a normal pair of glasses, but have a black device (telescope) protruding from the top of one lens for better identifying distance objects. The spectacle magnifier is mounted in a pair of glasses also for near vision

DETAILED DESCRIPTION:
You will be asked a series of oral questions regarding your health status and vision level of functioning (Expectations of Visual Functioning Form, NEI-VFQ, Linear Rating Scale, and Geriatric Depression Scale) in the Vanderbilt Eye Clinic. You will undergo a mobility pre-test to assess your ability to find objects in the distance as well as read . You will undergo a low vision examination in the eye clinic. You will receive the optical devices and then receive brief instructions on the use of the devices . You will then undergo a pre-training evaluation. You will receive approximately 6 training sessions with your prescribed devices for up to 1 hour each time. You will return to the Vanderbilt Eye Clinic for the post-training distance and near vision assessments with the devices . You will be asked the series of oral questions again regarding your health status and vision level of functioning .

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients with vision less than 20/40

Exclusion criteria:

- Subjects must not have any significant physical mobility limitations and be willing to participate in the testing and training sessions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-10; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
mobility | At time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Joos, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States